CLINICAL TRIAL: NCT01675986
Title: Comparing the Efficacy of Pregabalin and Hydroxyzine on the Anxiety Score
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GABAPAC
Record Dates: First submitted 2012-02-07; First posted 2012-08-30 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Feeling Anxious
MeSH Terms: conditions — Anxiety Disorders | interventions — Hydroxyzine; Pregabalin; Lactose

ARMS (3):
- Pregabaline (Experimental): Groups PREGABALINE : 150 mg de LYRICA®
  Interventions: Drug: Pregabalin
- Hydroxyzine (Experimental): Groups HYDROXYZINE : 75 mg d'ATARAX®
  Interventions: Drug: hydroxyzine
- Lactose (Placebo Comparator): Groups placebo : 4 g de lactose
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: hydroxyzine — 75 mg
  Arms: Hydroxyzine
Drug: Pregabalin — 150 mg
  Arms: Pregabaline
Drug: Lactose — 4 g
  Arms: Lactose

SUMMARY:
The insertion of long-lasting intravenous device is done under local anesthesia. Currently, in the investigators hospital, no premedication is given to the patients. However, this procedure occurs in a particular emotional context related to the diagnosis of cancer or malign hemopathies.

Therefore, administration of a sedative or anxiolytic drugs before the start of the procedure can be questionable.

Hydroxyzine is the reference molecule for premedication because of its anxiolytic and anti-histaminic properties A new agent, pregabalin, shares also the same properties

The main objective of this study was to compare the efficacy of pregabalin and hydroxyzine on the anxiety score as a premedication during the insertion of long-lasting intravenous device under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 75 years
* Patient schedules for insertion of long-lasting intravenous device

Exclusion Criteria:

* History of previous insertion of long-lasting intravenous device or central intravenous catheter
* long term treatment of gabapentin or pregabalin
* Hypersensitivity to pregabalin or any of the excipients
* Hypersensitivity to hydroxyzine, one of its metabolites, one of the excipients, another derivative of piperazine, aminophylline or ethylene diamine.
* Patient at risk of glaucoma e
* Patient at risk for urinary retention
* Patient severe respiratory failure
* Patient at the general condition not too corrupted (ASA IV)
* Renal failure with creatinin clearance < 30 ml / min
* Patient not affiliated to Social Security
* Pregnant or lactating
* Patients in emergency situations
* Inpatient without consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy treatment
  anxiety score VAS: 0 to 100

SECONDARY OUTCOMES:
Efficacy of pregabaldin
  anxiety score VAS:0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DEBAENE, MD, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU de POITIERS, Poitiers, France